CLINICAL TRIAL: NCT04506827
Title: Maxillary Sinus Augmentation With Three Different Biomaterials: Histologic, Histomorphometric, Clinical and Patient Reported Outcomes From a Randomized Controlled Trial
Brief Title: RCT With 3 Different Biomaterials for Maxillary Sinus Lift
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Antonio Barone, Professor, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SinusAug
Record Dates: First submitted 2020-07-22; First posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Alveolar Bone Atrophy
Keywords: Bone regeneration; Biomaterial(s); Implantology; Osseointegration
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Sinus Floor Augmentation

STUDY DESIGN:
Intervention Model Description: Three groups of patients will be treated with 3 different graft materials
Who Masked: Participant, Outcomes Assessor
Masking Description: The envelope with the group assignment will be opened by the surgeon at the time of surgery and the patient won't be informed.
  The clinician who registers clinical parameters won't be informed of the group allocation. The histologist will receive biopsies with a numeric code but without informations of the graft material used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (Active Comparator): patients in the control group received Demineralized Bovine Bone Mineral for the maxillary sinus augmentation
  Interventions: Procedure: Maxillary Sinus Augmentation; Device: Maxillary Sinus Graft with ABBM
- Test group 1 (Experimental): patients in the test group 1 received TCP with particle size from 250 to 1000 µm
  Interventions: Procedure: Maxillary Sinus Augmentation; Device: Maxillary Sinus Graft with TCP
- Test group 2 (Experimental): patients in the test group 2 received TCP as in test group1 plus crosslinked Hyaluronic Acid
  Interventions: Procedure: Maxillary Sinus Augmentation; Device: Maxillary Sinus Graft with TCP + HA

INTERVENTIONS:
Procedure: Maxillary Sinus Augmentation — Biomaterial Graft into the Maxillary Sinus
Device: Maxillary Sinus Graft with ABBM — The maxillary sinuses in the control group are grafted with ABBM
  Other Names: Anorganic Bovine Bone Mineral (ABBM)
  Arms: Control group
Device: Maxillary Sinus Graft with TCP — The maxillary sinuses in the test1 group are grafted with TCP
  Other Names: Tricalcium Phosphate (TCP)
  Arms: Test group 1
Device: Maxillary Sinus Graft with TCP + HA — The maxillary sinuses in the test1 group are grafted with TCP + HA
  Other Names: hyaluronic acid (HA)
  Arms: Test group 2

SUMMARY:
Background: Lateral maxillary sinus augmentation (MSA) is a predictable bone regeneration technique in case of atrophy of the posterior-upper maxilla. Aimed at obtaining quantity and quality of bone suitable for receiving osseointegrated implants, its success is largely due to the skill of the surgeon, but also to the characteristics of the biomaterial used.

Methods: Twenty-four patients needing MSA were included in the study. The patients were randomly allocated to 3 different groups: Anorganic Bovine Bone Mineral (ABBM) as control, Tricalcium Phosphate (TCP) with or without hyaluronic acid (HA) as test groups. Nine months after MSA bone biopsies were harvested for the histomorphometric analysis. Secondary outcomes were mean bone gain, intraoperative and post-operative complications, implant insertion torque, implant failure and patient related outcome measures (PROMs).

DETAILED DESCRIPTION:
The implant-prosthetic rehabilitation of the atrophic maxilla requires the creation of sufficient volumetric quantity of bone, through regeneration techniques, necessary to position the implants.

Maxillary sinus augmentation (MSA) is probably the most predictable and best performing technique.

The present randomized controlled study aims to evaluate and compare, histomorphometrically and clinically three different bone substitutes such as: ABBM, Tricalcium Phosphate (TCP) with or without the addition of hyaluronic acid (HA) that were used for lateral MSA. This study population will be followed until the 3rd year. This study describes histological differences between the three groups at 9 months.

All the patients enrolled in the study received a session of oral hygiene and a periodontal examination before the surgical procedure to obtain a more favorable oral environment for wound healing. A CBCT was mandatory for all included cases to verify that the maxillary sinus was clear and that the residual bone height was 3 mm or less. All the enrolled patients received 2 gr. of amoxicillin and clavulanic acid (or 600 mg. of clindamycin for those who were allergic to penicillins) as a pre-medication one-hour before surgery. All patients rinsed for 1 minute with 0.2% chlorhexidine mouthwash (and twice a day for the following 3 weeks). Local anesthesia was administered, a mid-crestal incision with mesial and distal release were performed to access the lateral bone wall of the maxillary sinus, subsequently, ultrasound bone surgery (Piezosurgery ®, Carasco, Italy) with specific tips was used for the bone window osteotomy (Figure 1-A). The Schneiderian membrane was reflected and lifted up medially with flat sinus curettes. Once the sinus membrane was completely lifted a bioabsorbable pericardium membrane (Smartbrane, Regedent AG, Zurich, Switzerland) was applied to protect it (Figure 1-B). The randomization sealed envelopes were opened and the clinician allocated the patients to one of the three experimental groups:

1. Control group that received Demineralized Bovine Bone Mineral (Bio-Oss Cancellous, Geistlich, Wolhunsen, Switzerland);
2. Test group 1 that received TCP with particle size ranging from 250 to 1000 µm (Osopia, Regedent, Zurich, Switzerland);
3. Test group 2 that received TCP as in test group1 plus crosslinked Hyaluronic Acid (Hyadent BG, Regedent, Zurich, Switzerland) with a ratio 2 to 1.

the bony window was repositioned, stabilized and covered with a resorbable pericardium membrane. Nine months after the MSA a CBCT analysis was required to evaluate the total bone height gain.

Depending on the treatment plan, between one and three implants, bone level (BL) or tissue level (TL), of two different manufacturers (Institut Straumann AG, Basel, Switzerland and Sweden & Martina, Due Carrare, Italy) were positioned. While preparing the osteotomy implant site a bone biopsy was harvested using a trephine. The implant insertion torque was measured in Ncm for each implant.

All patients were prescribed 1gr amoxicillin + clavulanic acid twice daily for 7 days (for those who were allergic to penicillin 300mg clindamycin 3 times daily for 7 days) as post-operative prophylaxis. All patients received 8mg of dexamethasone immediately after surgery and 4 mg of dexamethasone per day were prescribed for the following 5 days. Analgesics were prescribed (1gr paracetamol 3 times daily) according to patients' need. The use of removable temporary restorations was not recommended during the healing period.

After an osseointegration period of 3 months, the implants were restored. The prosthetic procedures were similar for all groups, impressions were taken with a polyether rubber material (Impregum, Espe Dental AG, Seefeld, Germany) and a customized impression tray. Final Zirconia screw-retained restorations were delivered after a period of 2/3 weeks, peri-apical radiographs were taken and oral hygiene instructions were given to all participants in the study.

ELIGIBILITY:
Inclusion Criteria:

* need for maxillary sinus augmentation
* 18 years or older
* residual ridge height less than 3mm

Exclusion Criteria:

* full contraindication to implant surgery,
* systemic diseases that could negatively influence wound healing;
* heavy smokers (more than 10 cigarettes/day);
* head and neck irradiation treatment;
* uncontrolled diabetes;
* chronic or acute sinus pathology;
* uncontrolled periodontal disease;
* full mouth plaque and bleeding score higher than 25%,
* tooth extractions in the previous 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2019-06-29 (Actual); Study Completion 2019-12-14 (Actual)

PRIMARY OUTCOMES:
Histomorphometric parameters of the augmented bone (descriptive) | 9 months
  Descriptive analysis of the specimen section at the microscope
Histomorphometric parameters of the augmented bone (% of new bone, marrow, graft) | 9 months
  Percentages of newly formed bone, marrow spaces and residual graft particles are reported.

SECONDARY OUTCOMES:
Mean bone gain measured at 9 months through CBCT evaluation | 9 months
  radiographic evaluation
Intra-operative | During surgery
  clinical evaluation (yes/no) of the presence or occurrence of: sinus membrane perforation, excessive bleeding, lateral sinus cortical bone fracture.
Post-operative complications | one week
  clinical evaluation (yes/no) of the presence or occurrence of:symptoms of acute sinusitis, swelling, suppuration, bleeding, trismus, hematoma, wound dehiscence, acute infections.
Post-operative complications | 9 months
  clinical evaluation (yes/no) of the presence or occurrence of:symptoms of chronic sinusitis, swelling, suppuration, wound dehiscence, acute infections.
Implant insertion torque measured in Ncm | 9 months
  clinical evaluation
Early implant failure | 12 months
  clinical evaluation of the osseointegration of the implant into the bone (yes/no)
Patient reported outcome measures | 9 months
  All patients will answer a questionnaire regarding the oral health-related quality of life using the 14 questions of the short-form Oral Health Impact Profile (OHIP-14) (This questionnaire consists of 14 questions each one formulated in the following way: "How often (impact item) because of problems with your teeth, mouth or dentures?" The impact items belong to 7 different impact domains: 1. Functional limitations; 2. Physical pain; 3. Psychological discomfort; 4. Physical disability; 5. Psychological disability; 6. Social disability; 7. Handicap. Each question can be answered with a score from 0 to 4 corresponding to: 0 = never, 1 = hardly ever, 2 = occasionally, 3 = fairly often, and 4 = very often.)

CONTACTS AND LOCATIONS:
Overall Officials: Nicola A Valente, DDS, MS, Study Chair — University of Seville, Spain
Locations (1):
- University of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No